CLINICAL TRIAL: NCT06975579
Title: A Study of the COherence of Scatter Identification and Exclusion Algorithm: The COSIE Study
Brief Title: The COherence of Scatter Identification and Exclusion Algorithm Study
Acronym: COSIE
Status: Recruiting | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Imperial College London (Other); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 5912; 24/NW/0086 (Other: NHS REC reference)
Record Dates: First submitted 2025-05-02; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Steatohepatitis, Nonalcoholic
Keywords: Liver ultrasound; backscatter coefficient; Non-alcoholic fatty liver disease; steatosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Staff at Royal Marsden Hospital or Institute of Cancer Research
  Interventions: Device: Ultrasound image processing
- Patients: Patients undergoing therapy/follow up for cancer with some evidence of non-alcoholic fatty liver disease.
  Interventions: Device: Ultrasound image processing

INTERVENTIONS:
Device: Ultrasound image processing — The COSIE study examines the coherence of ultrasound to improve the estimation of the backscatter coefficient.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is currently the most common liver condition worldwide; approximately 55% of the world population will have NAFLD by 2040. NAFLD is an unwanted side effect of common cancer therapies, such as chemotherapy. Ultrasound can detect NAFLD via measurement of the backscatter coefficient (BSC). It is an attractive technique because of its low cost and availability, potentially enabling earlier detection of NAFLD in a larger population through screening. This approach has shown promise in detecting NAFLD but is limited by variability in measurement due to several factors. Measurement of the BSC requires assumptions about the nature of the tissue being measured; if these assumptions are incorrect, they can lead to inaccurate BSC measurements. To improve accuracy, an algorithm (COSIE) was developed to quantify the suitability of tissue for BSC analysis. The investigators believe COSIE will enable more reliable BSC measurements by selecting the optimal regions of tissue to measure. By measuring the BSC in the livers of healthy volunteers and patients with evidence of fatty liver, the algorithm can be evaluated against liver fat percentage values obtained from MRI imaging. This study will assess whether applying the COSIE algorithm enhances the reliability of BSC measurements, bringing them closer in quality to MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Healthy male or female adults (18 or above).
* Volunteers must consider themselves fit and healthy.
* RMH and/or ICR employees.

Patients:

* Patients undergoing liver MRI as part of clinical standard of care with evidence of steatosis on preceding MRI.
* Aged 18 and above.

Exclusion Criteria:

Healthy Volunteers:

* Volunteers that are under investigation or planning to consult their GP to seek investigation for an undiagnosed condition, particularly regarding pelvic or abdominal disease or injury.
* Healthy volunteers who do not have an NHS number or who are not registered with a GP will be excluded.

Patients:

• Severe liver fibrosis (fibrosis stage F4) or severe cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is assumed that these volunteers will display a range of liver fat fractions and that there may be bias towards the low-fat fractions (< 5%). Patients with known fatty liver are included to present a broader range of cases to consider, thereby improving the analysis. If a patient is MR scanned and it is found that they have low fat fraction, we will aim to replace them with another patient that does have a high fat fraction.
  This number has been selected without a priori predictions of the expected variance in results. This study will help to determine the necessary study power required for future investigations. This population size has been selected based on practical considerations, i.e. cost of MR and length of the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Difference in backscatter coefficient | up to 6 months
  Mean difference in repeat measures of backscatter coefficient (BSC) in the liver with and without application of COSIE, across all participants and all views.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised ultrasound and MR images will be shared upon request.